CLINICAL TRIAL: NCT05984355
Title: Acceptability, Representations and Experiences of an Application Which Help the Walk for Older Persons
Brief Title: Acceptability, Representations and Experiences of an Application and Captors Which Suggest a Walking Itinerary
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Saint Etienne School of Mine (Other); Senior Autonomie (Unknown)
Responsible Party: Principal Investigator, Nathalie BARTH, PhD, Centre Hospitalier Universitaire de Saint Etienne
Other Study IDs: GA-2021-05
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Aging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- People aged 65 and over
  Interventions: Other: Individual interviews
- Naturals caregivers
  Interventions: Other: Individual interviews
- Professionals
  Interventions: Other: Individual interviews

INTERVENTIONS:
Other: Individual interviews — Discussion between the searcher and the participant about representations and acceptability about a potential application and captors which suggest a Walking itinerary

SUMMARY:
ParcourSenior is a project lead by School of Mines from Saint-Etienne, Gérontopôle AURA and "Senior Autonomie" to promote walking in a city environment. To enable that, we have two tools at your disposable. The first one is sensor which can measure physicals abilities. The second one is an application which proposes individual itineraries based on physical abilities. This application concern people whom want to walk alone, with supportive people or with new people encounter in this app. Both tools are in the process of being created. The current study focuses on needs, expectations and desire of the elders and professionals about both of these tools. After, we plan to focus on the acceptability of these devices. A qualitative study with focus groups is carried out to evaluate the needs and expectation follows by individual interviews to evaluate the project: acceptability, fears and use's perception.

DETAILED DESCRIPTION:
This research tend to study the acceptability of an application and captors which can propose a Walking itinerary of older 65 people.

ELIGIBILITY:
Inclusion Criteria:

* For first group : people aged 65 and over
* For natural caregivers : people who help in daily life a close relative
* For Professional : people who work with older person

Exclusion Criteria:

* Person with a neurological disease
* Person under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * person 65 years of age and older
  * natural caregivers
  * profesionnal who work with person 65 years of age and older
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
representations and acceptability about a potential application and captors which suggest a Walking itinerary | Days:30
  measure by individuals interviews

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Barth, PhD, Study Director — Gerontopole Auvergne Rhône Alpes
Locations (1):
- Gérontopole AURA, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No